CLINICAL TRIAL: NCT04982328
Title: Th17 Immune Response in Patients With COVID-19 and Nonalcoholic Fatty Liver Disease
Brief Title: COVID-19 and Nonalcoholic Fatty Liver Disease
Acronym: CovidFAT
Status: Completed | Type: Observational
Sponsor: University Hospital for Infectious Diseases, Croatia (Other)
Responsible Party: Sponsor
Other Study IDs: UHID07
Record Dates: First submitted 2021-07-24; First posted 2021-07-29 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Covid19; NAFLD
MeSH Terms: conditions — COVID-19; Non-alcoholic Fatty Liver Disease | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samples for cytokine analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NAFLD: patients diagnosed with NAFLD and hospitalized due to the severe COVID-19
  Interventions: Diagnostic Test: Th17 cytokine profile; Diagnostic Test: Screening for the components of metabolic syndrome; Diagnostic Test: Evaluation of the degree of steatosis
- non-NAFLD: patients hospitalized due to the with severe COVID-19 without NAFLD
  Interventions: Diagnostic Test: Th17 cytokine profile; Diagnostic Test: Screening for the components of metabolic syndrome; Diagnostic Test: Evaluation of the degree of steatosis

INTERVENTIONS:
Diagnostic Test: Th17 cytokine profile — Screening for the components of metabolic syndrome
Diagnostic Test: Screening for the components of metabolic syndrome — Anthropometric measures including height, weight, waist circumference and hip circumference will be measured in all patients. Results of the routine laboratory tests as part of the standard diagnostic procedure will be collected: CRP, leukocyte count, ratio neutrophils and lymphocytes, hemoglobin, platelet count, urea, creatinine, bilirubin, AST, ALT, GGT, ALP, albumins, fasting glucose.
Diagnostic Test: Evaluation of the degree of steatosis — The degree of steatosis will be estimated using the ultrasound and a method for grading steatosis will be measuring the degree of ultrasound attenuation by hepatic fat using a process based on simultaneous transient elastography (TE) which measures the degree of steatosis.

SUMMARY:
COVID-19 is currently the leading public health problem, associated with a high risk of complications and death in risk groups of patients. Non-alcoholic fatty liver disease (NAFLD) is the most common liver disease with a prevalence of 30% in the Western population and is also recognized as an independent risk factor for the development of severe COVID-19. In the pathogenesis of COVID-19, the key role is played by the hyperreactivity of the immune response, the so-called cytokine storm leading to the development of severe forms of pneumonia, acute respiratory and multiorgan failure. The aim of this study is to investigate the clinical course, outcomes, and profile of inflammatory response in patients with COVID-19 and NAFLD.

DETAILED DESCRIPTION:
SARS-CoV-2 virus infection is currently the leading public health problem, associated with a high risk of complications and death in at-risk groups. Risk factors for the development of severe forms of COVID-19 include components of the metabolic syndrome (obesity, diabetes, dyslipidemia, and arterial hypertension), which are also associated with the development of nonalcoholic fatty liver disease (NAFLD). According to previously published, but mostly retrospective studies, NAFLD is a possible risk factor for the development of severe COVID-19. . In the pathogenesis of COVID-19, the key role is played by the hyperreactivity of the immune response, the so-called cytokine storm. According to recent research, activation of the Th17 system could play a key role in the regulation of this excessive inflammatory response. Furthermore, Th17 lymphocytes and cytokines are important in the development and progression of NAFLD. The question is whether, due to Th17 hyperreactivity, patients with NAFLD are at higher risk of developing severe forms of the disease and what is the profile of the Th17 immune response to SARS-CoV-2 infection in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with COVID-19

Exclusion Criteria:

* Immunosuppression
* Consumption of alcohol > 20 g/day
* HIV
* Chronic viral hepatitis
* Presence of other chronic liver disease (hemochromatosis, Wilson's disease, toxic hepatitis, deficiency of alpha-1-antitrypsin, liver autoimmune disease)
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 120 patients diagnosed with and hospitalized for severe COVID-19 (60 patients with NAFLD, 60 patients without NAFLD).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Th17 cytokines concentrations | Day of hospital admission
  Measurement of Th17 cytokines concentration in serum of patients by multiplex technology

SECONDARY OUTCOMES:
Staging of liver steatosis | Day of hospital discharge (expected maximum of 28 days)
  The degree of steatosis will be estimated using the controlled attenuation parameter (CAP) in patients with NAFLD.
Duration of hospitalization | Day of hospital discharge (expected maximum of 28 days)
  Days of hospitalization
Remission of respiratory symptoms | Day of hospital discharge (expected maximum of 28 days)
  Time to independence from oxygen therapy in days
28 days survival | Day of hospital discharge (expected maximum of 28 days)
  Number of subjects surviving at 28 days from hospitalization
Rate of high flow oxygen therapy or non-invasive ventilation | Day of hospital discharge (expected maximum of 28 days)
  Requirement for high flow oxygen therapy during the initial hospitalisation
Secondary infections | Day of hospital discharge (expected maximum of 28 days)
  Presence/absence of secondary infection during hospitalization
Rate of invasive mechanical ventilation | Day of hospital discharge (expected maximum of 28 days)
  Requirement of invasive mechanical ventilation
Rate of pulmonary thromboembolism | Day of hospital discharge (expected maximum of 28 days)
  Presence of pulmonary thromboembolism diagnosed with MSCT pulmonary angiography on clinical suspicion

CONTACTS AND LOCATIONS:
Overall Officials: Neven Papic, MD, PhD, Principal Investigator — School of Medicine, University of Zagreb, Croatia
Locations (1):
- University Hospital for Infectious Diseases Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mocibob L, Susak F, Situm M, Viskovic K, Papic N, Vince A. COVID-19 and Pulmonary Thrombosis-An Unresolved Clinical Puzzle: A Single-Center Cohort Study. J Clin Med. 2022 Nov 29;11(23):7049. doi: 10.3390/jcm11237049. PMID 36498623
- [Result] Papic N, Samadan L, Vrsaljko N, Radmanic L, Jelicic K, Simicic P, Svoboda P, Lepej SZ, Vince A. Distinct Cytokine Profiles in Severe COVID-19 and Non-Alcoholic Fatty Liver Disease. Life (Basel). 2022 May 26;12(6):795. doi: 10.3390/life12060795. PMID 35743825
- [Result] Susak F, Vrsaljko N, Vince A, Papic N. TGF Beta as a Prognostic Biomarker of COVID-19 Severity in Patients with NAFLD-A Prospective Case-Control Study. Microorganisms. 2023 Jun 13;11(6):1571. doi: 10.3390/microorganisms11061571. PMID 37375073
- [Result] Vrsaljko N, Samadan L, Viskovic K, Mehmedovic A, Budimir J, Vince A, Papic N. Association of Nonalcoholic Fatty Liver Disease With COVID-19 Severity and Pulmonary Thrombosis: CovidFAT, a Prospective, Observational Cohort Study. Open Forum Infect Dis. 2022 Feb 9;9(4):ofac073. doi: 10.1093/ofid/ofac073. eCollection 2022 Apr. PMID 35287335